CLINICAL TRIAL: NCT02213705
Title: Treatment of Refractory Sever Systemic Scleroderma by Injection of Allogeneic Mesenchymal Stem Cells
Acronym: MSC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC Severe Systemic Sclerosis
Record Dates: First submitted 2014-07-17; First posted 2014-08-11 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2020-10

CONDITIONS: SYSTEMIC SCLERODERMA; ALLOGENEIC MESENCHYMAL STEM CELLS; ADULT
Keywords: SYSTEMIC SCLERODERMA; TRANSPLANTATION; ALLOGENEIC MESENCHYMAL STEM CELLS; ADULT
MeSH Terms: conditions — Scleroderma, Systemic

ARMS (1):
- INJECTION OF ALLOGENEIC MESENCHYMAL STEM CELLS (Experimental): Administration of allogeneic MSCs in the treatment of severe diffuse SSc or rapidly progressive and refractory to conventional treatments by prior cyclophosphamide
  Interventions: Biological: INJECTION OF ALLOGENEIC MESENCHYMAL STEM CELLS

INTERVENTIONS:
Biological: INJECTION OF ALLOGENEIC MESENCHYMAL STEM CELLS

SUMMARY:
The main ailm of this phase I-II study is to evaluate toxicity and efficacy of allogenic mesenchymal stem cell therapy to treat severe systemic sclerosis. In practice this treatment will be given to patients with a rapidly evolutive disease or refractory to cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years and <70 years.
* Established diagnosis of systemic sclerosis according to the criteria of the American College of Rheumatology
* SSc of poor prognosis, involving life-threatening with sever visceral impairment (cardiac, pulmonary or renal) AND " a) contraindicating the use of or b) resistant to " immunosuppressive therapy conventionally used in severe forms of the disease according to the European recommendations of EUSTAR (www.eustar.org) and EBMT (www.ebmt.org) which then rely on high doses of iv cyclophosphamide (either in monthly bolus at least six months or by intensification and autograft of Hematopoietic Stem Cells) or SSc with fibrosing lung damage threatening the vital prognosis which excludes a lung transplant.

These forms of severe and serious SSc WITH at least 6 months follow-up after completion of prior immunosuppressive therapy by high doses of iv cyclophosphamide when they were made, combine to varying degrees : rapidly progressive skin lesions with a score of Rodnan> 15 and one or more of the major visceral lesions defined as follows :

1. Respiratory disease :

   DLCO <60% or FVC ≤70% of the theoretical value and the presence of interstitial lung disease (abnormalities on chest radiograph and / or lung HRCT with thin sections). It is necessary to ensure that non-related etiologies to scleroderma were eliminated; example: obstructive lung disease (chronic obstructive pulmonary disease or pulmonary emphysema). If the fibrosing lung disease threatens the vital prognosis, we will ensure of the exclusion of a possible lung transplant.

   And/or
2. Heart disease:

congestive heart failure reversible, ventricular or atrial rhythm disturbances defined as recurrent episodes of atrial fibrillation or atrial flutter, recurrent paroxysmal atrial tachycardia or ventricular tachycardia, atrioventricular block of second or third degree, pericardial effusion with high abundance needing specific treatment of medical type (introduction of steroids) or surgical type (drainage). It is necessary to ensure that non-related etiologies to scleroderma were removed.

* Signed informed consent.
* Presence of a consenting intrafamilial MSC donor
* Affiliation to social security.

Exclusion Criteria:

* Pregnancy or absence of appropriate contraception throughout the study.
* Respiratory Disease:
* systolic Pulmonary arterial pressure (PASP)>55mmHg (on echocardiography or after right heart catheterization);
* DLCO <30% of the theorical ;
* Respiratory failure defined by oxygen arterial pressure at rest (PaO2) <8 kPa (<60 mmHg) and / or a blood pressure of carbon dioxide at rest (PaCO2)> 6.7 kPa (> 50 mmHg) without oxygen therapy.

Renal Disease:

* Calculated creatinine clearance <20 ml/mn/m2
* Sequelae cystopathy post treatment by cyclophosphamide
* Heart disease:
* Clinical sign of a congestive heart failure refractory ;
* Left ventricular ejection fraction <35% at myocardial scintigraphy or echocardiography;
* Pulmonary arterial hypertension confirmed by right catheterization or suspected pulmonary hypertension with systolic PAP at echography > 40 mmHg
* Chronic atrial fibrillation requiring oral anticoagulant therapy;
* Uncontrolled ventricular arrhythmia;
* Pericardial effusion with hemodynamic compromise assessed by echocardiography.
* Hepatic Disease:
* Hepatic impairment defined as a persistent increase in transaminases or bilirubin to 3 times normal.
* Psychiatric disorders, including drug taking and alcohol abuse.
* Active neoplasia or concomitant myelodysplasia, antecedent of neoplasia.
* Bone marrow failure defined by neutropenia <0.5 x 109 / L, thrombocytopenia <50 x 109 / L, anemia <8 g / dL, CD4 lymphopenia <200 x 106 / L.
* Uncontrolled systemic hypertension.
* Uncontrolled acute or chronic infection, HIV1, 2 or HTLV-1, 2seropositivity.
* Chronic hepatitis B or C active.
* Significant exposure to bleomycin, toxic oils, vinyl chloride, trichloroethylene or silica; eosinophilia-myalgia syndrome, eosinophilia fasciitis.
* Risk of poor patient compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05-06 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Immediate Toxicity | 10 days
  Immediate Toxicity/tolerance defined as grade 3 or above toxicity base on the CTCAE - Cancer Therapy Evaluation Program (CTEP), observed during the first 10 days (http://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/ctcaev3.pdf)

SECONDARY OUTCOMES:
Medium-term tolerance | 2 years
  Treatment-related event-free survival at 2 years. Treatment-related event (morbidity) being defined by the onset of clinical events induced by the procedure and not explained by the natural or expected course of the scleroderma disease.
Survival | 2 years
  Time from inclusion to death
Progression free survival | 2 years
  Defined as the time in days from the day of inclusion until the occurrence of changes compared to the initial assessment, documented and re-evaluated at two successive examinations 3 months
CBC | 1, 2, 3, 4, 8, 12, 16, 20, 24 weeks
  complete blood count (CBC)
Platelet | 1, 2, 3, 4, 8, 12, 16, 20, 24 weeks
  Platelet blood count
Lymphocyte | 3, 6, 9, 12, 15, 18, 24 months
  Lymphocyte subpopulation blood count measured by flow cytometry
Antibody | 3, 6, 9, 12, 15, 18, 24 months
  Antibody response
Rodnan score | 3, 6, 9, 12, 15, 18, 24 months
  modified Rodnan Score
SHAQ | 3, 6, 9, 12, 15, 18, 24 months
  Scleroderma Health Assessment Questionnaire (SHAQ)
Clinical progression | 3, 6, 9, 12, 15, 18, 24 months
  Occurence of visceral involvement, defined as any of the following:
  * Pulmonary: diffusion capacity of CO (DLCO and DLCO/VA), forced vital capacity (FVC), total lung capacity (TLC), residual volume (RV), pulmonary artery pressure (measured by echocardiography or right heart catheterisation), arterial blood gases (pO2, pCO2, p(A-a)O2) in ambient air,
  * Myocardial: ECG, left ventricular function measured by echocardiography (and cardiac MRI and/or Gating in the event of cardiac abnormality or suspected LV dysfunction on ultrasound) with semi-quantitative analysis of the degree of cardiac damage according to the cardiac score (based on the presence or absence of left axial deviation on the electrocardiogram and/or moderate or significant pericardial effusion according to the echocardiogram),
  * Renal: 24-hour proteinuria, creatinine clearance,
  * Patient's weight in kg,
Clinical response | 3, 6, 9, 12, 15, 18, 24 months
  Defined by a 25% improvement in modified Rodnan Score and/or ≥10% in DLCO or FVC compared to baseline state without the need to reintroduce other immunosuppressants.

CONTACTS AND LOCATIONS:
Overall Officials: dominique farges, MDPHD, Principal Investigator — APHP
Locations (1):
- Saint-Louis Hospital, Paris, France

REFERENCES:
- [Background] Farge D, Loisel S, Resche-Rigon M, Lansiaux P, Colmegna I, Langlais D, Charles C, Pugnet G, Maria ATJ, Chatelus E, Martin T, Hachulla E, Kheav VD, Lambert NC, Wang H, Michonneau D, Martinaud C, Sensebe L, Cras A, Tarte K. Safety and preliminary efficacy of allogeneic bone marrow-derived multipotent mesenchymal stromal cells for systemic sclerosis: a single-centre, open-label, dose-escalation, proof-of-concept, phase 1/2 study. Lancet Rheumatol. 2022 Feb;4(2):e91-e104. doi: 10.1016/S2665-9913(21)00326-X. Epub 2022 Jan 5. PMID 38288741
- [Derived] Loisel S, Lansiaux P, Rossille D, Menard C, Dulong J, Monvoisin C, Bescher N, Bezier I, Latour M, Cras A, Farge D, Tarte K. Regulatory B Cells Contribute to the Clinical Response After Bone Marrow-Derived Mesenchymal Stromal Cell Infusion in Patients With Systemic Sclerosis. Stem Cells Transl Med. 2023 Apr 17;12(4):194-206. doi: 10.1093/stcltm/szad010. PMID 36928395